CLINICAL TRIAL: NCT06480513
Title: The Effect of Yoga on Endocrine Therapy Induced Musculoskeletal Symptoms in Women With Breast Cancer: the COBRA Study
Brief Title: Cancer Of the BReast Asanas Study (COBRA)
Acronym: COBRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: World Cancer Research Fund International (Other)
Responsible Party: Principal Investigator, Dr. Evelyn Moninkhof, Assistant professor, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-054/G; NL86325.041.24
Record Dates: First submitted 2024-06-12; First posted 2024-06-28 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga group (Experimental): following live yoga classes twice a week and using yoga video's at home once a week
  Interventions: Behavioral: live yoga
- control group (Other): Waiting list control group. The control group will be offered live remote yoga classes after the intervention period
  Interventions: Behavioral: live remote yoga

INTERVENTIONS:
Behavioral: live yoga — following live yoga classes twice a week and using yoga video's at home once a week
  Arms: yoga group
Behavioral: live remote yoga — The control group will be offered live remote yoga classes after the intervention period
  Arms: control group

SUMMARY:
Rationale: Women with hormone-receptor positive breast cancer are usually prescribed endocrine therapy for a period of 5-10 years. This treatment reduces the risk of recurrence and improves overall survival in these women. Musculoskeletal complaints are a common (~50%) negative consequence of endocrine treatment, which affects daily functioning and quality of life. These symptoms frequently result in early treatment discontinuation, which is associated with shorter disease-free survival. Musculoskeletal complaints are often pharmacologically treated with limited effect and accompanied by side-effects. Therefore, interventions to counteract musculoskeletal complaints are urgently needed in this population. A potential non-pharmacological option is yoga. In patients with osteoarthritis, there is emerging evidence that yoga is effective to reduce pain and stiffness and improve function. Yoga as treatment for musculoskeletal complaints that are associated with endocrine treatment is rarely investigated and mainly in small studies.

Objective: The objective of the proposed study is to assess the effectiveness of a 4-month yoga program compared to a waiting list control group on musculoskeletal complaints in women with hormone-positive stage I-III breast cancer receiving endocrine treatment who report musculoskeletal complaints.

Study design: The COBRA study is a randomized controlled trial with two study arms: a yoga- and a waiting list control group.

Study population: For this study, 140 women with oestrogen-receptor positive stage I-III breast cancer on endocrine treatment (aromatase inhibitors; >4 months) will be recruited. These women experience musculoskeletal complaints (>3 months) which started or exacerbated after initiation of endocrine treatment. Furthermore, eligible women did not practice yoga in the last six months and are not planning to start yoga and are not highly physically active (i.e., >150 minutes per week moderate-vigorous exercise).

Intervention: The intervention consists of two one-hour sessions/week supervised yoga and once a week 30-minute yoga exercises at home. The 4-month yoga program will be an active form of yoga, such as Easy Vinyasa yoga, which is characterized by continuous slow movements linked with breathing. The waiting list control patients will be offered an online yoga program after the 4-month study period.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with oestrogen-receptor positive stage I-III breast cancer,
* Use of aromatase inhibitors (>4 months and will continue using it for at least six months),
* Have finished primary treatment (chemotherapy, radiotherapy, surgery) for at least six weeks,
* Experience musculoskeletal complaints (>3 months, which are at least mild in severity (i.e., score of ≥ 3 for worst pain item of a modified version of the Brief Pain Inventory [BPI](16, 42))., which started or exacerbated after initiation of endocrine treatment,
* Be stabilized on menopausal symptom medication or antidepressants for at least three months and three weeks, respectively(19), if applicable, and
* Be able to read, speak and understand Dutch or English.

Exclusion Criteria:

* Too physically active (i.e., >150 minutes/week of self-reported moderate-to-vigorous or leisure and sports activities)
* Following (during the last 6 months), or planned to follow yoga classes on a structural base
* Following, or planned to follow, a structured psychological intervention during the intervention period, i.e., cognitive behavioral therapy, or unstable on psychotropic medication
* Participated in the intervention group of an exercise study during breast cancer treatment
* Any circumstances that would impede ability to give informed consent or adherence to study requirements as determined by the study team
* More than 2 weeks not able to attend training sessions during the intervention period

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal complaints | Baseline, at 4 and 8 months
  Worst of joint pain and stiffness/joint pain and stiffness severity/joint pain and stiffness interference assessed by the modified version of the BPI

SECONDARY OUTCOMES:
Lower extremity joint complaints | Baseline, at 4 and 8 months
  Using the WOMAC questionnaire
Upper extremity musculoskeletal complaints | Baseline, at 4 and 8 months
  Using the DASH questionnaire
Menopausal symptoms | Baseline, at 4 and 8 months
  Using the FACT-ES questionnaire
Fatigue | Baseline, at 4 and 8 months
  Using the MFI questionnaire
Sleep | Baseline, at 4 and 8 months
  Using the PSQI questionnaire
Quality of Life | Baseline, at 4 and 8 months
  Using the QLQ-C30 that has functional scales, symptom scales and a global quality of life (QOL) score. A high score for a functional scale represents a high/ healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of Life | Baseline, at 4 and 8 months
  Using the BR45. The QLQ-BR45 incorporates nine multi-item scales to assess body image, sexual functioning, breast satisfaction, systemic therapy side effects, arm symptoms, breast symptoms, endocrine therapy symptoms, skin mucosis symptoms, endocrine sexual symptoms. All items are scored 1 to 4.
Anxiety and depression | Baseline, at 4 and 8 months
  Using the Hospital Anxiety and Depression Scale (HADS) where anxiety and depression are measured separately on a scale from 0-7 (Normal), 8-10 (borderline abnormal) and 11-21 (abnormal).
Cognitive problems | Baseline and at 4 months
  Using the Amsterdam Cognition Scan
Cognitive problems | Baseline, at 4 and 8 months
  Using the FACT-COG
Habitual physical activity | Baseline, at 4 and 8 months
  Using the Short Questionnaire to Assess Health-enhancing physical activity (SQUASH). Physical activity is measured in minutes per week.
Blood markers | Baseline and at 4 months
  Inflammatory markers (Interleukin-6 and Interleukin-IB, tumor necrosis factor alpha (TNF-alpha) and high-sensitive C-reactive protein (hsCRP). At the end of the study we will conduct a literature review to identify the most promising biomarkers.
Physical strength | Baseline and at 4 months
  Hand grip strength using a handgrip dynamometer. The best of three attempts will be recorded.
Physical strength | Baseline and at 4 months
  Leg press using a hypothetical 1-RM test
Physical fitness | Baseline and at 4 months
  Steep ramp test using a cycle ergometer
Vital signs | Baseline and at 4 months
  Blood pressure and resting heart rate
Anthropometrics | Baseline and at 4 months
  Weight and height will be combined to report BMI in kg/m^2. Waist- and hip circumference.
Safety of the yoga intervention | 0-8 months (whole study period)
  (Serious) adverse events potentially related to the intervention
Use of pain medication | 0-8 months (whole study period)
  Self-reported with a diary
Compliance with endocrine treatment | 0-8 months (whole study period)
  Self-reported with a diary

CONTACTS AND LOCATIONS:
Overall Officials: Anne May, Prof. Dr., Study Director — UMC Utrecht
Locations (1):
- University Medical Center Utrecht (UMC Utrecht), Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided